CLINICAL TRIAL: NCT03881839
Title: Impact of "Internet Tools" Consultation on Increasing Emergency Attendance
Brief Title: Internet Tools and Emergency Attendance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-431; 2019 / CE 06 (Other: 2019 / CE 06)
Record Dates: First submitted 2019-03-07; First posted 2019-03-20 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Emergency
MeSH Terms: conditions — Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient in emergency department
  Interventions: Other: emergency

INTERVENTIONS:
Other: emergency — The objective of this research will be to assess, in patients presenting in an emergency department, the prior consultation of medical information on a website, the impact on the emergency consultation decision and the relevance of this consultation.

SUMMARY:
Over the years, there has been an increase in the flow of emergency rooms, which is gradually leading to an overcrowding of emergency unit. This overcrowding is multifactorial with, for example, a decrease in the outpatient care in family medicine and specialized medicine, emergency services unsuitable at the level of premises ... In parallel, investigator note in recent years facilitated access to internet and especially to GAFA which is the acronym for Google, Amazon, Facebook, Apple. As a result, patients have 24-hour access to medical information via websites, blogs and social networks. This information of, often, unreliable medical information can lead to ambiguity among patients about the need for urgent or delayed intervention in the management of their symptoms. In fact, "everything becomes urgent". To date, in France, no study has evaluated the impact and prevalence of consulting a website for medical purposes before consulting an emergency service. The objective of this research will be to assess, in patients presenting in an emergency department, the prior consultation of medical information on a website, the impact on the emergency consultation decision and the relevance of this consultation.

DETAILED DESCRIPTION:
It is an observational study, monocentric, prospective. This study consists in collecting data from an anonymized questioner given to patients presenting themselves at the emergency department of Clermont-Ferrand University Hospital. Answers to the questions will not change the patient's management. The questioner, containing 17 questions, requires answering "yes" or "no" by ticking boxes, or even specify when it is stipulated. This questionnaire will be given to the patient after his registration, and filled by the latter in the waiting room, pending medical care. Answering the questionnaire will take between 5 to 10 minutes. The data is anonymous.

The patient arrives at the emergency department and registers at the entrance desks where a paper and computer file is created. Then, the Reception and Orientation Nurse takes care of the patient by welcoming him in the reception box, she realizes the taking of the hemodynamics constants, the collection of the reason of consultation with the grievances of the patient. During this phase, patient will be inform of the completion of this study and asked to participate in this study. If the patient agrees to participate, an anonymized questioner will be provided and explained by one of the investigating physicians or associated partners.

ELIGIBILITY:
Inclusion Criteria:

* Any major patient presenting to the emergency department by their personal way.

Exclusion Criteria:

* Suspicion of acute alcoholism
* dementia
* guardianship / trusteeship
* language barrier, non-communicating patient
* patient refusing to participate in the study
* patient with confusion
* patient with Glasgow scale less than 15
* patient not affiliated with social security
* patient not knowing how to read or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any major patient presenting to the emergency department by their personal way.
Sampling Method: Non-Probability Sample
Enrollment: 431 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Rate of justified nature of the consultation between patient who did consult a website before the emergency room and those who didn't. | at day 1
  The comparison between the justification (or not) of the transition to adult emergencies and the consultation of an upstream website will be done using the Chi2 test (or Fisher's exact test if applicable).
  The search for criteria related to the justified nature of this emergency procedure will be done with the Chi2 test (or Fisher's exact test if applicable) for the categorical data and with the Student's test (or Mann and Whitney test if not normally distributed) for continuous data.

SECONDARY OUTCOMES:
Prevalence of Internet consultation among patients admitted to emergency room | at day 1
  The rate of consultation of a website before the emergency room, will be expressed as a percentage with its 95% confidence interval
The rate of justified consultation | at day 1
  The rate of justified consultation to emergency department, will be expressed as a percentage with its 95% confidence interval.
Risk factors related to consultation of a website medical information prior to the transition to adult emergencies. | at day 1
  The comparison between patients who visited a medical information website (vs those who did not consult the internet) before the emergency department visit will be done using the same methods as for the analysis of the main criterion.

CONTACTS AND LOCATIONS:
Overall Officials: Farès MOUSTAFA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France